CLINICAL TRIAL: NCT03058835
Title: IN-US-276-1340: Pre-Exposure Prophylaxis to Prevent HIV Acquisition in US Women: A Demonstration Project
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Shobha Swaminathan, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro20150001562; IN-US-276-1340 (Other: Gilead Sciences Inc.)
Record Dates: First submitted 2017-02-08; First posted 2017-02-23 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: PrEP Adherence Monitoring
Keywords: HIV; Truvada
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- PrEP with Truvada (Experimental): All study participants will be assigned to this arm and will receive Truvada tablets (tenofovir disoproxil and emtricitabine) for PrEP
  Interventions: Drug: tenofovir disoproxil and emtricitabine

INTERVENTIONS:
Drug: tenofovir disoproxil and emtricitabine — Pre-exposure Prophylaxis with Truvada will be distributed to all participants eligible to receive PrEP.
  Other Names: Truvada tablets

SUMMARY:
The overall aim of this study is to assess attitudes toward PrEP, feasibility of Truvada PrEP procurement through the established access procedures, and adherence to Truvada PrEP among US women at risk for HIV acquisition.

DETAILED DESCRIPTION:
Study Design:

This is a 24 week prospective pilot study assessing attitudes toward and feasibility of using Truvada PrEP in a population of women at risk for HIV acquisition.At this site 31 HIV- uninfected women desiring PrEP will be enrolled at each site (confirm number). We will have to consent about 50 women which includes screen failures.The study will assess attitudes towards and adherence to PrEP with questionnaires at weeks 12 and 24. Tenofovir levels procured at week 12 and 24 week of PrEP will be used to assess adherence to PrEP.

Primary objectives:

1. Describe attitudes toward PrEP among a population of women at risk for HIV acquisition, living in HIV prevalent areas.
2. Assess feasibility of Truvada procurement through the established Gilead access program
3. Evaluate adherence at week 12 and week 24 using dried blood spots

Secondary objective:

1. Describe HIV incidence
2. Describe associations of positive and negative attitudes toward PrEP with acceptance of PrEP and subsequent adherence
3. Assess adherence at weeks 12 and 24
4. Evaluate the relationship between PrEP adherence and sexual activity
5. Compare geographic areas with respect to PrEP attitudes
6. Mentor junior investigators at each site.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 64 years old
* Able to give consent
* "At risk" for HIV as defined by any of the following:

  1. unprotected sex (in past 6 months) with 1 or more men of unknown HIV status
  2. evaluated for an STI within 6 months prior to screening
  3. sex in last 6 months with an HIV-infected partner
  4. IDU with report of using previously used or shared needles in past 6 months or has been in a methadone, buprenorphine, or suboxone treatment program in past 6 months or engaging in high-risk sexual behaviors
  5. individuals engaging in transactional sex (i.e sex for money, drugs, or housing)
  6. Infrequently uses condoms during sex with 1 or more partners of unknown HIV status who are known to be at substantial risk of HIV infection (IDU or bisexual male partner)
* CrCl ≥ 60 ml/min
* HIV- uninfected women desiring PrEP

Exclusion Criteria:

* Active alcohol or drug use or dependence which may interfere with adherence to study requirements
* HIV-infected at screening or enrollment
* Estimated CrCl < 60 mL/min
* Past participation in an HIV vaccine study
* Positive Hepatitis B surface antigen test
* Underlying medical condition with survival unlikely during follow-up period
* Any condition that in the opinion of study staff would make participation in the study unsafe or interfere with achieving study objectives
* Pregnant or breast feeding
* Actively trying to achieve pregnancy

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 125 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Describe attitudes toward PrEP among a population of women at risk for HIV acquisition, living in HIV prevalent areas | 24 Weeks
  Attitudes towards PrEP will be assessed with questionnaires at weeks 12 and 24.
Assess feasibility of Truvada procurement through the established Gilead access program | 24 Weeks
  Logistic regression comparing the proportion of participants with tenofovir plasma levels greater than 0.3 will be analyzed
Evaluate adherence to Truvada PrEP at week 12 and week 24 using dried blood spots | 24 Weeks
  Adherence to Truvada PrEP will be assessed at week 12 and week 24 using dried blood spots and questionnaire responses concerning adherence to PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Shobha Swaminathan, MD, Principal Investigator — New Jersey Medical School
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - New Jersey Medical School Clinical Research Center, Newark, New Jersey
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT03058835/ICF_000.pdf